CLINICAL TRIAL: NCT04646473
Title: Thinking Outside the Clinic: A Digital Health Approach for Young Adults With Type 1 Diabetes
Brief Title: Sweetgoals for Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Catherine Stanger, Associate Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 23559; R01DK124428 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- App only (Experimental): Sweetgoals app only
  Interventions: Behavioral: SweetGoals app
- App plus Incentives (Experimental): SweetGoals app + incentives=yes + coaching=no
  Interventions: Behavioral: SweetGoals app; Behavioral: Incentives
- App plus Coaching (Experimental): Sweetgoals app + incentives=no + coaching=yes
  Interventions: Behavioral: SweetGoals app; Behavioral: Coaching
- App plus Coaching plus Incentives (Experimental): Sweetgoals app + incentives=yes + coaching=yes
  Interventions: Behavioral: SweetGoals app; Behavioral: Coaching; Behavioral: Incentives

INTERVENTIONS:
Behavioral: SweetGoals app — App offers goal setting and feedback
Behavioral: Coaching — Web health coaching
  Arms: App plus Coaching; App plus Coaching plus Incentives
Behavioral: Incentives — Financial incentives for meeting goals
  Arms: App plus Coaching plus Incentives; App plus Incentives

SUMMARY:
The study will test an app and web-delivered intervention designed to improve glycemic control (HbA1c) among young adults with Type 1 diabetes. All participants will receive the "core" digital intervention, the SweetGoals app, focused on self-monitoring and goal setting. Efficacy of two independent intervention components (incentives for adherence and web health coaching) will be tested

DETAILED DESCRIPTION:
ASSIGNMENT OF PARTICIPANTS:

Interested participants will download the SweetGoals app. Once all screening procedures are complete, including A1c verification via the mail in test kit, research staff will schedule a web video meeting to (1) randomize participants and inform them of their intervention condition assignment; (2)assist participants in setting up their Glooko account and uploading their devices and orient them to the Glooko data visualization hub; and (3) download the Glooko mobile app, which may be used by all participants and into which participants without a Glooko compatible pump will enter carb counts.

INTERVENTION DELIVERY:

All participants will receive the core intervention, the SweetGoals app. Those assigned to Incentives will receive the app plus incentives for meeting adherence goals. Those assigned to Coaching will receive web health coaching to increase motivation and skill in self-management as described below.

DIABETES CARE FOR ALL PARTICIPANTS:

Participants in all conditions will receive ongoing treatment for type 1 diabetes from their current medical provider. Report of a visit within the past 6 months is a study inclusion criterion. Study staff will not provide medical care or intervention. All participants will receive information about recommendations for medical care related to diabetes (e.g., quarterly visits and A1c assessment, consistent with Standards of Medical Care in Diabetes). Informational links will be provided within SweetGoals for various online resources addressing T1D educational topics.

CORE INTERVENTION FOR ALL PARTICIPANTS: SWEETGOALS APP

All participants will receive the SweetGoals app, an automated intervention that sets weekly self-management goals and provides weekly feedback. The SweetGoals app will be implemented and delivered using the MobileCoach app platform, which runs on both Android and iOS systems. The SweetGoals app sends weekly reminders to upload devices, retrieves device data via the Glooko API, applies decision rules to evaluate daily and weekly goals, and sends weekly feedback messages about goal adherence and encouragement about adherence in the upcoming week.

Diabetes Self-Management Goals. Glooko stores multiple variables that are used to evaluate the glucose monitoring and mealtime goals. Across both glucose monitoring and mealtime target behaviors, we use a similar structure to the goals to promote ease of remembering the goals and communication with participants. Specifically, regardless of the devices used or the target (glucose monitoring or mealtime behaviors) there is a daily adherence goal, and there is a weekly goal of meeting the daily goal on >5 days each week. These weekly goals were selected to promote high consistency in mealtime glucose monitoring and carb counting. Each week, participants will be asked to set personal goals for the next week for the number of days they think they can meet each daily goal. Each week they will receive a message stating the number of days on which they met each goal, how that compared to their personal goal, and whether they met the ultimate weekly goal (met daily goal >5 days per week).

Glucose monitoring goals. Each participant will receive a device-specific (glucometer vs. CGM) daily goal based on the device they use to monitoring their glucose levels, and the ultimate weekly goal for all participants is to meet the daily goal on at least 5 days per week. For participants who use a glucometer only, the daily self-monitoring of blood glucose (SMBG) goal is >5 checks, each >2 hours from another check. For participants who use CGM, the CGM wear time goal is 80% of expected values each day. Expected values per day are based on the device-specific check frequency (e.g., every 5 mins for Dexcom G6). We selected this cutoff to reflect clinically necessary glucose monitoring frequency, but also allow for legitimate disconnect time (sports, leisure activities) and sensor changes.

Mealtime goals. Each participant will receive daily goals specific to their insulin delivery method (pump vs. MDI). Participants will be asked to check their glucose before they eat (if they use a glucometer only, not CGM). Participants who use a Glooko compatible pump will only need to use their pump to document the mealtime goals. If they use a pump+glucometer combination that requires manual entry of the glucose value into the pump, they must complete the glucose check and that manual entry no longer than 30 minutes before the carb entry to receive credit for meeting the mealtime goal. If they use a pump+CGM or other meter that transfers the glucose value to the pump without manual entry, no manual entry is necessary. If they use MDI (no insulin pump), they will use the Food event screen to enter their carb counts in the Glooko smartphone app.

When each participant's Glooko data are retrieved, our algorithm evaluates whether or not there is a valid glucose value within 30 minutes prior to each carb entry. The daily mealtime target is 3 paired glucose level/carb count values.

INCENTIVE COMPONENT

In addition to using the SweetGoals app, participants assigned to Incentives will also receive incentives for meeting goals. Incentives to improve adherence to glucose monitoring and mealtime behaviors that support appropriate insulin bolusing are paid weekly from weeks 1-11, then fade in frequency from weeks 12-25, a procedure used to promote long lasting improvements in adherence and A1c. In the fading phase, incentives are paid at increasing time intervals (i.e., 2,3,4 then 5-week delays; paid at weeks 13, 16, 20, 25).

For meeting daily and weekly goals, participants can earn the following incentives: (1) $1 for each day meeting glucose monitoring goal. (maximum=$7 per week); (2) $5 per week bonus for meeting the glucose monitoring goal 6 or 7 days to promote consistent weekly glucose monitoring. (maximum=$5 per week) (3) $1 for every day with >3 properly timed glucose value/carb entry pairs (maximum=$7 per week); (4) $5 per week bonus for meeting the mealtime goal 6 or 7 days to promote consistent weekly glucose checking and carb counting at mealtime. (maximum=$5 per week). Total earnings possible each week are $24 (~$3.50 per day). The maximum earnings for all goals are $600 across 25 weeks. Research staff will load earned incentives on reloadable prepaid MasterCards.

WEB HEALTH COACHING COMPONENT:

Participants assigned to coaching will also receive 15 Web Health Coaching sessions by a bachelors-level health coach. These coaching sessions are designed to promote effective self-management of diabetes. Coaching sessions are held weekly from weeks 1-11, then fade over the second half of the intervention with 4 sessions held during weeks 12-25 (weeks 13, 16, 20, and 25). Sessions 1-7 are 30 minutes each, as new material is introduced and practiced. Sessions 8-15 are 15 minutes each, as problem solving skills are practiced and applied to new challenges identified by participants. Coaching will be completed using Zoom, an online HIPAA compliant web conference system.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of T1D for >18 months
* Have A1c ≥7.5%
* Report a visit with physician managing type 1 diabetes (T1D) within the previous 6 months
* Participants must use a glucometer or continuous glucose monitor compatible with Glooko.

Exclusion Criteria:

* Pregnancy or breast feeding
* Severe medical illness that would preclude participation (e.g., cystic fibrosis, developmental disability, severe cognitive impairment)
* Psychiatric illness that would preclude participation
* Diabetes diagnoses other than T1D (Type 2 Diabetes, Maturity Onset Diabetes of the Young/MODY)
* Use of any medications known to impact glycemic control (oral or injectable corticosteroids, beta-blockers, antipsychotic medications such as risperidone).
* A history of known hemoglobinopathy, anemia, or transfusion (which could alter the validity of HbA1c measurement)
* Already being engaged in a psychological intervention targeting diabetes adherence.

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | +12 months
  Mean HbA1c

SECONDARY OUTCOMES:
Glucose checking adherence | +12 months
  Mean proportion of days in the past 30 meeting daily glucose checking goal
Problem solving | +12 months
  Mean score on the Social Problem Solving Inventory-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Stanger, Ph.D., Principal Investigator — Trustees of Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers and practitioners, while safeguarding the privacy of participants and protecting confidential and proprietary data and third-party intellectual property. Findings will be published as soon as they are available in relevant peer-reviewed journals that are available online, and share as requested directly to the author(s). Data requests can be made directly to the Principal Investigator with information for accessing the data on the NIDDK Data Repository.
Supporting Information: Study Protocol
Time Frame: If the study ends and data are no longer being obtained directly from study participants by study investigators, all study data will be provided to the Repository by the end of the funding period (which may include no-cost extensions). The period of exclusive use of the entire dataset from the study will be for three years after the last study contact for collection of intervention outcomes.
Access Criteria: Data requests made directly to the Principal Investigator or through the NIDDK Data Repository

REFERENCES:
- [Derived] Plaitano EG, Stanger C. Joint effect of nicotine use and diabetes distress on glycemic control in young adults with type 1 diabetes. J Diabetes Complications. 2025 Aug;39(8):109083. doi: 10.1016/j.jdiacomp.2025.109083. Epub 2025 May 17. PMID 40398346
- [Derived] Stanger C, Kowatsch T, Xie H, Nahum-Shani I, Lim-Liberty F, Anderson M, Santhanam P, Kaden S, Rosenberg B. A Digital Health Intervention (SweetGoals) for Young Adults With Type 1 Diabetes: Protocol for a Factorial Randomized Trial. JMIR Res Protoc. 2021 Feb 23;10(2):e27109. doi: 10.2196/27109. PMID 33620330